CLINICAL TRIAL: NCT02878837
Title: Dex vs Dazzle: Dexmedetomidine vs Midazolam for Intraoperative Sedation
Brief Title: Dexmedetomidine vs Midazolam for Intraoperative Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo (Other)
Responsible Party: Principal Investigator, João manoel Silva Junior, Director, Department of Anesthesiology, Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAMSPE
Record Dates: First submitted 2016-08-10; First posted 2016-08-25 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Failed Moderate Sedation During Procedure; Minimally Conscious State
MeSH Terms: conditions — Persistent Vegetative State | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DEX (Active Comparator): Patients undergoing surgical procedures under regional anesthesia sedated with a loading dose of 1 µg/Kg of Dexmedetomidine over 10 minutes followed by continuous infusion at 0.2 to 0.8 µg/Kg/h, along with 0.5µg/Kg bolus breakthrough doses of Fentanyl as necessary to achieve a RASS score between -3 and -1.
  Interventions: Drug: Dexmedetomidine
- MDZ (Active Comparator): Patients undergoing surgical procedures under regional anesthesia sedated with a 0.05mg/Kg bolus dose of Midazolam, along with 0.02 mg/Kg bolus doses of Midazolam plus 0.5µg/Kg bolus doses of Fentanyl as necessary to achieve a RASS score between -3 and -1
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: DEX
Drug: Midazolam
  Arms: MDZ

SUMMARY:
This randomized, open clinical trial sought to compare the use of Midazolam and Dexmedetomidine during surgery in patients under regional anesthesia.

The primary objective was to determine the superiority of either drug during the intraoperative period regarding: 1- Depth of sedation and 2- incidence of complications.

Secondary objectives included the determination of superiority regarding the postoperative period.

For that, patients were randomized into two groups and sedated with either Midazolam or Dexmedetomidine.

DETAILED DESCRIPTION:
This study was a randomized, open clinical trial.

Patients undergoing surgery under regional (neuraxial or brachial plexus block) anesthesia were randomly assigned into one of two groups.

Patients in one of the groups (called MDZ) were initially sedated with a 0.05mg/Kg bolus dose of Midazolam.

The ones in the other group (called DEX) were initially sedated with a loading dose of 1 µg/Kg of Dexmedetomidine over 10 minutes, followed by continuous infusion at 0.2 to 0.8 µg/Kg/h.

In order to achieve a Richmond Agitation-Sedation Scale (RASS) score between -3 and -1, the following breakthrough doses were used as necessary:

MDZ: 0.02 mg/Kg bolus dose of Midazolam plus 0.5µg/Kg bolus dose of Fentanyl DEX: 0.5µg/Kg bolus dose of Fentanyl

Depth of sedation and incidence of complications were recorded during surgery, in the Post Anesthesia Care Unit (PACU) and in the Ward for two days following surgery,

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery under regional anesthesia

Exclusion Criteria:

* The presence of any Bradyarrhythmia;
* New York Heart Association (NYHA) Functional Classes III and IV Heart Failure and/or Left Ventricle Ejection Fraction under 30%;
* Respiratory Failure, Glasgow Coma Scale score 8 or under, and Liver Failure - due to the increased risk of sedation in patients with these conditions (d) refusal to participate in the study or withdrawal of consent at any moment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Depth of Sedation | Intraoperative
  Number of breakthrough doses necessary to achieve RASS score between -3 and -1
Respiratory depression | Intraoperative
  Use of supplemental oxygen flow greater than 2L/min or endotracheal intubation for mechanical ventilation
Bradycardia | Intraoperative
  Heart Rate < 50 heartbeats per minute
Hypotension | Intraoperative
  Mean Arterial Pressure < 55mmHg

SECONDARY OUTCOMES:
Residual Sedation | Up to 2 hours after surgery
  RASS score < -1 in Post Anesthesia Care Unit
Shivering | Up to 2 hours after end of surgery
  Self-described by the patient
Pain | 2 days
  Pain, described by the patient, according to the Analog Scale. Necessity of breakthrough doses of analgesics.
Quality of Sleep | 2 days
  Self-described.
Delirium | 2 days
  Incidence of Delirium according to CAM-ICU algorithm
Length of Hospital Stay | Until Discharge, up to 30 days
  Length of time between surgery and discharge from Hospital, in days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital do Servidor Publico Estadual, São Paulo, Sao Paulo SP, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostermann ME, Keenan SP, Seiferling RA, Sibbald WJ. Sedation in the intensive care unit: a systematic review. JAMA. 2000 Mar 15;283(11):1451-9. doi: 10.1001/jama.283.11.1451. PMID 10732935
- [Background] Bailey PL, Pace NL, Ashburn MA, Moll JW, East KA, Stanley TH. Frequent hypoxemia and apnea after sedation with midazolam and fentanyl. Anesthesiology. 1990 Nov;73(5):826-30. doi: 10.1097/00000542-199011000-00005. PMID 2122773
- [Background] American Society of Anesthesiologists Task Force on Sedation and Analgesia by Non-Anesthesiologists. Practice guidelines for sedation and analgesia by non-anesthesiologists. Anesthesiology. 2002 Apr;96(4):1004-17. doi: 10.1097/00000542-200204000-00031. No abstract available. PMID 11964611
- [Background] Candiotti KA, Bergese SD, Bokesch PM, Feldman MA, Wisemandle W, Bekker AY; MAC Study Group. Monitored anesthesia care with dexmedetomidine: a prospective, randomized, double-blind, multicenter trial. Anesth Analg. 2010 Jan 1;110(1):47-56. doi: 10.1213/ane.0b013e3181ae0856. Epub 2009 Aug 27. PMID 19713256
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Background] Ebert TJ, Hall JE, Barney JA, Uhrich TD, Colinco MD. The effects of increasing plasma concentrations of dexmedetomidine in humans. Anesthesiology. 2000 Aug;93(2):382-94. doi: 10.1097/00000542-200008000-00016. PMID 10910487
- [Background] Venn RM, Hell J, Grounds RM. Respiratory effects of dexmedetomidine in the surgical patient requiring intensive care. Crit Care. 2000;4(5):302-8. doi: 10.1186/cc712. Epub 2000 Jul 31. PMID 11056756
- [Background] Arain SR, Ebert TJ. The efficacy, side effects, and recovery characteristics of dexmedetomidine versus propofol when used for intraoperative sedation. Anesth Analg. 2002 Aug;95(2):461-6, table of contents. doi: 10.1097/00000539-200208000-00042. PMID 12145072
- [Background] Venn RM, Grounds RM. Comparison between dexmedetomidine and propofol for sedation in the intensive care unit: patient and clinician perceptions. Br J Anaesth. 2001 Nov;87(5):684-90. doi: 10.1093/bja/87.5.684. PMID 11878517
- [Background] Elbaradie S, El Mahalawy FH, Solyman AH. Dexmedetomidine vs. propofol for short-term sedation of postoperative mechanically ventilated patients. J Egypt Natl Canc Inst. 2004 Sep;16(3):153-8. PMID 15959548
- [Background] Abdalla MI, Al Mansouri F, Bener A. Dexmedetomidine during local anesthesia. J Anesth. 2006;20(1):54-6. doi: 10.1007/s00540-005-0351-z. PMID 16421680
- [Background] Taghinia AH, Shapiro FE, Slavin SA. Dexmedetomidine in aesthetic facial surgery: improving anesthetic safety and efficacy. Plast Reconstr Surg. 2008 Jan;121(1):269-276. doi: 10.1097/01.prs.0000293867.05857.90. PMID 18176230
- [Background] Usta B, Gozdemir M, Demircioglu RI, Muslu B, Sert H, Yaldiz A. Dexmedetomidine for the prevention of shivering during spinal anesthesia. Clinics (Sao Paulo). 2011;66(7):1187-91. doi: 10.1590/s1807-59322011000700011. PMID 21876972
- [Background] Bajwa SJ, Gupta S, Kaur J, Singh A, Parmar S. Reduction in the incidence of shivering with perioperative dexmedetomidine: A randomized prospective study. J Anaesthesiol Clin Pharmacol. 2012 Jan;28(1):86-91. doi: 10.4103/0970-9185.92452. PMID 22345953
- [Background] Belleville JP, Ward DS, Bloor BC, Maze M. Effects of intravenous dexmedetomidine in humans. I. Sedation, ventilation, and metabolic rate. Anesthesiology. 1992 Dec;77(6):1125-33. doi: 10.1097/00000542-199212000-00013. PMID 1361310
- [Background] Takrouri MS, Seraj MA, Channa AB, el-Dawlatly AA, Thallage A, Riad W, Khalaf M. Dexmedetomidine in intensive care unit: a study of hemodynamic changes. Middle East J Anaesthesiol. 2002 Oct;16(6):587-95. PMID 12503262
- [Result] Gertler R, Brown HC, Mitchell DH, Silvius EN. Dexmedetomidine: a novel sedative-analgesic agent. Proc (Bayl Univ Med Cent). 2001 Jan;14(1):13-21. doi: 10.1080/08998280.2001.11927725. PMID 16369581
- [Result] Gerlach AT, Murphy CV. Dexmedetomidine-associated bradycardia progressing to pulseless electrical activity: case report and review of the literature. Pharmacotherapy. 2009 Dec;29(12):1492. doi: 10.1592/phco.29.12.1492. PMID 19947809
- [Result] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Result] Tan JA, Ho KM. Use of dexmedetomidine as a sedative and analgesic agent in critically ill adult patients: a meta-analysis. Intensive Care Med. 2010 Jun;36(6):926-39. doi: 10.1007/s00134-010-1877-6. Epub 2010 Apr 8. PMID 20376429
- [Result] Chrysostomou C, Schmitt CG. Dexmedetomidine: sedation, analgesia and beyond. Expert Opin Drug Metab Toxicol. 2008 May;4(5):619-27. doi: 10.1517/17425255.4.5.619. PMID 18484919
- [Result] Grosu I, Lavand'homme P. Use of dexmedetomidine for pain control. F1000 Med Rep. 2010 Dec 17;2:90. doi: 10.3410/M2-90. PMID 21283652
- [Result] Kettner SC, Willschke H, Marhofer P. Does regional anaesthesia really improve outcome? Br J Anaesth. 2011 Dec;107 Suppl 1:i90-5. doi: 10.1093/bja/aer340. PMID 22156274
- [Result] Shir Y, Raja SN, Frank SM. The effect of epidural versus general anesthesia on postoperative pain and analgesic requirements in patients undergoing radical prostatectomy. Anesthesiology. 1994 Jan;80(1):49-56. doi: 10.1097/00000542-199401000-00011. PMID 8291729
- [Result] Huupponen E, Maksimow A, Lapinlampi P, Sarkela M, Saastamoinen A, Snapir A, Scheinin H, Scheinin M, Merilainen P, Himanen SL, Jaaskelainen S. Electroencephalogram spindle activity during dexmedetomidine sedation and physiological sleep. Acta Anaesthesiol Scand. 2008 Feb;52(2):289-94. doi: 10.1111/j.1399-6576.2007.01537.x. Epub 2007 Nov 14. PMID 18005372
- [Result] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Derived] Silva-Jr JM, Katayama HT, Nogueira FAM, Moura TB, Alves TL, de Oliveira BW. Comparison of dexmedetomidine and benzodiazepine for intraoperative sedation in elderly patients: a randomized clinical trial. Reg Anesth Pain Med. 2019 Mar;44(3):319-324. doi: 10.1136/rapm-2018-100120. Epub 2019 Feb 3. PMID 30777901